CLINICAL TRIAL: NCT04555265
Title: Investigation of Cytokine Change and Its Prognostic Value in Patients With Hepatocellular Carcinoma Treated by Thermal Ablation
Brief Title: Cytokine Change in Hepatocellular Carcinoma Treated by Thermal Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Society of Gastroenterology (Unknown)
Responsible Party: Principal Investigator, Kelvin K.C. Ng, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001kkcng/surg/cuhk
Record Dates: First submitted 2020-09-11; First posted 2020-09-18 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: cytokine; hepatocellular; carcinoma; thermal; ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Patients with hepatocellular carcinoma treated by thermal ablation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thermal ablation group (Other): Patients with hepatocellular carcinoma treated by thermal ablation
  Interventions: Device: Radiofrequency ablation or microwave ablation

INTERVENTIONS:
Device: Radiofrequency ablation or microwave ablation — Hepatocellular carcinoma treated by either radiofrequency ablation or microwave ablation

SUMMARY:
Background: Hepatocellular carcinoma (HCC) is the most common primary liver cancer with aggressive tumor behavior. Radiofrequency ablation (RFA) or microwave ablation (MWA) is an effective curative treatment for early stage HCC. This thermal ablation of liver tumor induces host immune response with changes in serum concentration of various cytokines. It is not clear whether this host immune response correlates with tumor recurrence and long-term patient survival.

Objective: This prospective study is to investigate the change of cytokines' level following RFA or MWA for HCC and its clinical correlation with tumor recurrence and patients' long-term survival data.

Hypothesis: Thermal ablation of HCC creates tumor antigen source for the generation of antitumor immunity and enhances host immune responses. The resulting inflammation and changes in cytokines may augment tumor cell death by increasing neutrophil infiltration and oxidative burst mechanisms. On the other hand, there may be negative effects via the production of growth factors, which could stimulate tumor cell growth within the sub-lethal margin. Therefore, the ultimate clinical consequences would be significantly affected by these immune responses.

Study design: This is a prospective study on the measurement of changes of serum cytokines in patients with HCC undergone RFA or MWA using the commercially available kit (MILLIPEX, Human cytokine/chemokine magnetic bead panel - Immunology Multiplex Assay ), which measure 10 cytokines, including IL-1β, IL-6, IL-10, IL-12 (p40), IL-12 (p70), TNF-α, CXCL8, CXCL9, CXCL10, CCL2, CCL5. Statistical correlation will be performed between the cytokine change and long-term patients' clinical outcome using the prospectively collected database.

Subjects: Patients with HCC undergone RFA or MWA in the Department of Surgery, The Chinese University of Hong Kong will be recruited. Exclusion criteria were evidence of extrahepatic metastasis, patients receiving combined hepatectomy and other local ablative therapy and patients with decompensated liver function that preclude local ablative treatment.

Intervention: RFA or MWA will be performed for patients with HCC. The serum samples of all consecutive recruited patients will be collected prospectively during the intervention. The measurement of cytokines level will be performed in the Laboratory of Department of Chemical Pathology, The Chinese University of Hong Kong under the standard protocol.

Main outcome measures: Primary outcome measure is early intrahepatic tumor recurrence within one year after thermal ablation. Secondary outcome measures are other tumor recurrence pattern (late intrahepatic recurrence and extrahepatic metastasis), overall survival and recurrence-free survival.

Data analysis: All data will be prospectively collected by a research assistant and computerized in a database. Statistical analysis will be performed by Chi-square test or Fisher's exact test, where appropriate, to compare discrete variables and Mann-Whitney U test to compare continuous variables. Cumulative survival will be computed by the Kaplan-Meier method and compared by Log-rank test. Multivariable analysis using logistic regression model will be done to identify the independent prognostic factors affecting early tumor recurrence.

Expected results: Understanding the relationship between the cytokines change during thermal ablation and post-treatment tumor recurrence helps to identify high risk patients for the possible adjuvant therapy in future study.

DETAILED DESCRIPTION:
Background Liver cancer is the sixth most common malignancy in the world. It is the fourth leading cause of cancer-related deaths and has a global incidence of more than 840,000 new cases in 2018.1 Hepatocellular carcinoma (HCC) accounts for 75% - 85% of primary liver cancer. Hepatectomy, radiofrequency ablation (RFA) and orthotopic liver transplantation are the main treatment options for patients with early stage HCC.2 Hepatectomy is only indicated in patients with early stage HCC and preserved liver function, whereas the application of liver transplantation is limited globally because of organ shortage. RFA is therefore the most effective treatment in patients with HCC and borderline liver function due to cirrhotic liver, especially in Asia-Pacific region where hepatitis B infection is prevalent.

Thermal ablation kills tumors via direct thermal denaturation and coagulation of tumor proteins.3 The retention of devitalized and damaged tumor cells within the body stimulates a robust inflammatory response. It has also been reported that thermal ablation creates a tumor antigen source for the generation of antitumor immunity and enhances host immune responses.4 Activated platelets release interleukin (IL) -1, tumor necrosis factor (TNF), and transforming growth factor , which increase vascular permeability and promote chemotaxis. Neutrophils are attracted to the ablation site and perform debris scavenging by releasing free radicals via oxidative burst mechanisms aimed at destroying inciting agents. Macrophage migration ensues, transitioning to the proliferative stage, during which macrophages secrete growth factors, including TNF, vascular endothelial growth factor (VEGF) and basic fibroblast growth factor.5 The level of proliferative activity of macrophages and lymphocytes is mediated by IL-6 positively and IL-10 negatively.6, 7 In the event of an incomplete ablation or nearly complete ablation, viable tumor cells in the sub-lethal ablation zone) may be affected positively or negatively by the concomitant inflammatory response including increased levels of cytokines and growth factors. Inflammation following ablation may have negative effects via the production of growth factors and cytokines by macrophages and lymphocytes, which could stimulate tumor cell growth within the sub-lethal zone.8 Human and animal studies using immunohistochemical staining of tissues, enzyme-linked immunosorbent assay of tissue lysates, and enzyme-linked immunosorbent assay of plasma have shown significant increase in specific inflammatory and immunomodulatory mediators after RFA.9, 10 The principle investigator has previously reported the inflammatory responses of RFA using the porcine liver model that the level of systemic inflammatory markers (TNF and IL-1) was significantly elevated after RFA, when compared with hepatectomy.11 Although pre-clinical studies on inflammatory responses of thermal ablation for liver tumor are substantial, clinical correlation of these micro-environmental reaction is limited in the literature. Erinjeri et al.12 reported that the ablation type and primary diagnosis predicted the change of IL-6 and patient age predicted the change of IL-10 after thermal ablation of tumors. IL-6 may act as surrogates for immunogenic cell death and the combination of immunogenic death-inducing procedures with immune check-point inhibitor may be beneficial to prolong patient survival after RFA.13 At the cellular level, RFA has proven to enhance tumor-associated antigen-specific T cell response and this contributes to the HCC recurrence-free survival of patients.14 Nonetheless, it is still not clear about the possible relationship between RFA-induced cytokines change and its prognostic value on tumor recurrence and long-term patient survival.

The principle investigator has reported the results of 209 patients receiving RFA as the sole treatment for HCC.15 The overall tumor recurrence rate was up to 80% with median follow-up of 26 months. Hence, identification of high-risk patients who might develop early recurrence using surrogate biomarkers (e.g. cytokines) carries an important clinical implication on the use of adjuvant treatment (e.g. immune check-point inhibitor).

Therefore, the investigators propose this single-center prospective study to analysis the change in serum cytokines level in patients with HCC treated by RFA or MWA. The result will be used to correlate the clinical outcome of patients, especially tumor recurrence and long-term survival outcome. This proposed clinical trial is of clinical importance in establishing the potential role of immune response as surrogate biomarkers to predict long-term patient outcome. It establishes the platform for future study of adjuvant treatment using immune check-point inhibitor for patients with HCC treated by RFA or other thermal ablative therapy. The investigators' center is a tertiary referral center in Hong Kong managing patients with complicated hepatobiliary and pancreatic diseases. The number of new cases of patients with HCC managed in the investigators' center is around 200 every year and the number of patients with HCC undergoing hepatectomy is around 80 every year. All the investigators are experts with vast experience in clinical and basic researches of patients with HCC. The investigators have conducted and published several randomized trials on management of HCC and other aspects of hepatobiliary surgery in international journals.16-19

Hypothesis RFA or MWA for HCC might induce inflammatory immune response with resulting change in cytokines level. This micro-environmental reaction might positively or negatively regulate the residual tumor cells, leading to the significant changes in tumor recurrence and long-term patient survival.

Aim of study This prospective study aims to investigate the change of cytokines' level following RFA or MWA for HCC and its clinical correlation with tumor recurrence and patients' long-term survival data. Primary outcome measure is early tumor recurrence within one year after RFA. Secondary outcome measures are other tumor recurrence pattern (late intrahepatic recurrence and extrahepatic metastasis), overall survival and recurrence-free survival.

Primary outcome measure is early intrahepatic tumor recurrence within one year after RFA and MWA. Secondary outcome measures are other tumor recurrence pattern (late intrahepatic recurrence and extrahepatic metastasis), overall survival and recurrence-free survival.

Analysis of cytokines level using studied patient serum samples

Analytes available:

IL-1β, IL-6, IL-10, IL-12 (p40), IL-12 (p70), TNF-α, CXCL8, CXCL9, CXCL10, CCL2, CCL5

Commercially available kit:

MILLIPLEX MAP Human Cytokine/Chemokine Magnetic Bead Panel - Immunology Multiplex Assay

Application of kit:

Simultaneously analyze multiple cytokine and chemokine biomarkers with MILLIPLEX MAP Human Cytokine/Chemokine Magnetic Bead Panel - Immunology Multiplex Assay, in human serum, plasma and cell culture samples. This is an overnight incubation assay.

Expected time of study The investigators' institution is a major tertiary referral center for HCC in Hong Kong. The patient recruitment will be started once the approval from Institution Review Board is obtained. The recruitment period is around 12 months to 18 months. With the median follow-up period of around 18 months, It is expected that the total period of study is three years.

Sample size estimation Expected number of patients to be recruited is estimated at 60 according to the past patient number undergoing treatment under the department.

Statistical analysis All data will be prospectively collected by a research assistant and computerized in a database. Statistical analysis will be performed by Chi-square test or Fisher's exact test, where appropriate, to compare discrete variables and Mann-Whitney U test to compare continuous variables. Cumulative survival will be computed by the Kaplan-Meier method and compared by Log-rank test. Multivariable analysis using logistic regression model will be done to identify the independent prognostic factors affecting early tumor recurrence.

Ethical Consideration This study will be carried out in accordance with the Declaration of Helsinki of the World Medical Association and the International Conference on Harmonization - Good Clinical Practice.

Consent Written voluntary consent will be obtained after full explanation of the trial to the patient before operation and randomization.

Relevance to clinical applications

This study carries significant clinical influence on the surgical management of patient with HCC. Since hepatitis B infection is still endemic in Asia-Pacific area like Hong Kong, hepatitis B related HCC is still a burden among the whole pool of cancer patients. This study aims to establish the potential role of immune response as surrogate biomarkers to predict long-term patient outcome. It enhances the development of the platform for future study of adjuvant treatment using immune check-point inhibitor for patients with HCC treated by thermal ablative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with HCC undergoing RFA or MWA will be recruited into this study provided the following criteria are fulfilled.

  1. HCC of maximal diameter < 8cm, and/or
  2. Multiple tumor nodules < 5, and/or
  3. Normal liver (serum total bilirubin level < 50 umol/L and serum albumin > 30 g/L) and renal function (serum creatinine level <120 mmol/L)
  4. Child-Pugh class A or B

Exclusion Criteria:

1. Evidence of extrahepatic metastasis
2. Patients receiving combined hepatectomy and other local ablative therapy
3. Patients with decompensated liver function that preclude local ablative treatment.
4. Patients with previous treatment for HCC (TACE, radiofrequency ablation, high intensity focus ultrasound or systemic chemotherapy)
5. Patients with inadequate serum sample for cytokine analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Early tumor recurrence | 12 months
  Early intrahepatic tumor recurrence within one year after RFA and MWA

SECONDARY OUTCOMES:
Other tutor recurrence | up to 24 months
  Late intrahepatic recurrence and extrahepatic metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No